CLINICAL TRIAL: NCT02716610
Title: Samba-02: An Investigation of the Dose-Response and Subject Variability of Inhaled Insulin in Subjects With Type 2 Diabetes
Brief Title: Dose-Response and Variability of Inhaled Insulin in Type 2 Diabetes
Acronym: Samba-02
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dance Biopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Samba-02
Record Dates: First submitted 2016-03-09; First posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- INH 69 U (low) (Experimental): single 69 U dose administration of Dance inhaled human insulin using a low-concentration formulation (300 U/mL)
  Interventions: Drug: INH 69 U (low)
- INH 69 U (high) (Experimental): single 69 U dose administration of Dance inhaled human insulin using a high-concentration formulation (900 U/mL)
  Interventions: Drug: INH 69 U (high)
- INH 139 U (Experimental): single 139 U dose administration of Dance inhaled human insulin using a high-concentration formulation (900 U/mL) This arm was repeated in order to evaluate intra-subject variability.
  Interventions: Drug: INH 139 U
- INH 208 U (Experimental): single 208 U dose administration of Dance inhaled human insulin using a high-concentration formulation (900 U/mL)
  Interventions: Drug: INH 208 U
- LIS 18 U (Active Comparator): single 18 U dose administration of subcutaneous insulin lispro using a 100 U/mL formulation This arm was repeated in order to evaluate intra-subject variability.
  Interventions: Drug: LIS 18 U

INTERVENTIONS:
Drug: INH 69 U (low) — inhaled human insulin
  Other Names: Dance-501
  Arms: INH 69 U (low)
Drug: INH 69 U (high) — inhaled human insulin
  Other Names: Dance-501
  Arms: INH 69 U (high)
Drug: INH 139 U — inhaled human insulin
  Other Names: Dance-501
  Arms: INH 139 U
Drug: INH 208 U — inhaled human insulin
  Other Names: Dance-501
  Arms: INH 208 U
Drug: LIS 18 U — subcutaneous insulin lispro
  Other Names: subcutaneous insulin lispro
  Arms: LIS 18 U

SUMMARY:
Pharmacokinetic (PK) and Pharmacodynamic (PD) dose-response investigation of Dance-501 inhaled human insulin

DETAILED DESCRIPTION:
This study investigated the pharmacokinetic (PK) and pharmacodynamic (PD) properties of Dance-501, a novel inhaled human insulin liquid formulation (INH) and device. Twenty-four subjects with type 2 diabetes (T2DM) received 3 INH doses: low (69 units), medium (139 units) and high (208 units) and 1 equivalent medium dose (18 units) of subcutaneous insulin lispro (LIS).

The medium dose was repeated to determine within subject variability. PD was investigated during a 12 hour euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus treated with insulin injections at a total daily dose less than 1.2 U/kg/day.
* Body mass index 25-40 kg/m2
* Hemoglobin A1c 6.5-9.5%
* Forced vital capacity and forced expiratory volume in 1 second at least 75% of predicted normal values.
* Fasting c-peptide less than 1 nmol/L

Exclusion Criteria:

* Any condition possibly affecting drug absorption from the lung, in particular subjects with decreased lung function or subjects taking bronchodilators or subjects who smoke.
* Active or chronic pulmonary disease.
* Any major disorder other than type 2 diabetes.
* Decompensated heart failure or myocardial infarction at any time or angina pectoris within the last 12 months.
* Proliferative retinopathy or maculopathy or severe neuropathy.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve for insulin from 0-8 hours (AUCins0-8h) | 0 to 8 hours following each dose
  Assessment of the linearity of the dose-response curves
Maximum concentration of insulin (CMaxIns) | up to 12 hours following each dose
  Assessment of the linearity of the dose-response curves
Area under the curve for glucose infusion rate from 0-12 hours (AUGgir0-12h) | 0 to 8 hours following each dose
  Assessment of the linearity of the dose-response curves
Maximum glucose infusion rate (GIRmax) | up to 12 hours following each dose
  Assessment of the linearity of the dose-response curves

SECONDARY OUTCOMES:
Bioavailability | 0 to 8 hours following each dose
  Relative delivery efficiency (FREL) of inhaled human insulin (INH) compared to subcutaneous injected insulin lispro (LIS)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH

IPD SHARING:
Plan to Share IPD: No